CLINICAL TRIAL: NCT05480579
Title: A Dose Escalation Phase I Clinical Study to Evaluate the Tolerability and Safety of a Single Intravenous Injection IBI311 in Healthy Volunteers
Brief Title: A Study of IBI311 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI311A101
Record Dates: First submitted 2022-07-15; First posted 2022-07-29 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: treated with different doses of single intravenous injection of IBI311 (Experimental)
  Interventions: Biological: IBI311
- Cohort 1: placebo group (Placebo Comparator)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: placebo — Dose4 placebo of single IV injection
  Arms: Cohort 1: placebo group
Biological: IBI311 — Dose2 IBI311 of single IV injection
  Arms: Cohort 1: treated with different doses of single intravenous injection of IBI311
Biological: IBI311 — Dose4 IBI311 of single IV injection
  Arms: Cohort 1: treated with different doses of single intravenous injection of IBI311
Biological: placebo — Dose3 placebo of single IV injection
  Arms: Cohort 1: placebo group
Biological: placebo — Dose1 placebo of single IV injection
  Arms: Cohort 1: placebo group
Biological: IBI311 — Dose1 IBI311 of single IV injection
  Arms: Cohort 1: treated with different doses of single intravenous injection of IBI311
Biological: IBI311 — Dose 3 IBI311 of single IV injection
  Arms: Cohort 1: treated with different doses of single intravenous injection of IBI311
Biological: placebo — Dose2 placebo of single IV injection
  Arms: Cohort 1: placebo group

SUMMARY:
It is designed for Multi-center, double-masked, randomized, placebo- control study with dose escalation phase I trial to evaluate the safety, tolerability, PK and immunogenicity profiles of a single intravenous injection of IBI311 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to sign informed consent form and comply with visit and study procedures per protocol.
2. Male or female subjects with age of 18~45 yrs.
3. Female subjects of childbearing age or male subjects with childbearing age female partner agree to take effective contraceptive measures from the screening period to 120 days after the end of treatment.

Exclusion Criteria:

1. Have a history of or any evidence of chronic diseases of liver, kidney, cardiovascular, nervous/mental, digestive tract, respiratory, urinary and endocrine systems.
2. Have received prior treatment with another anti-IGF-1R monoclonal antibody.
3. History of drug, alcohol, or chemical abuse within 6 months prior to screening.
4. History of positive HIV antibody, HCV antibody, Syphilis check, HBV positive during screening period.
5. Receipt of a live vaccine within 180 days prior to screening or expected to receive live vaccine during study period.
6. History of recurrent significant infection or history of recurrent bacterial infections.
7. Must not have a history of tinnitus or hearing impairment.
8. Must not have received an investigational agent for any condition within 90 days.
9. Female volunteers must not be pregnant or lactating.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
Incidence, relatedness and severity of all adverse events, treatment emergent adverse events and serious adverse events | Up to 16 weeks

SECONDARY OUTCOMES:
maximum concentration (Cmax） | Up to 16 weeks.
  PK parameters maximum concentration (Cmax） of IBI311
area under the curve (AUC) | Up to 16 weeks.
  PK parameters area under the curve (AUC) of IBI311
half-life (t1/2) | Up to 16 weeks.
  PK parameters half-life (t1/2) of IBI311
the incidence of ADA | Up to 16 weeks
  Positive rate of anti-drug antibody

CONTACTS AND LOCATIONS:
Overall Officials: Yongfang Yuan, Ph D., Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No